CLINICAL TRIAL: NCT06366412
Title: Effect of Dexmedetomidine on Serum Tau-217 Protein as a Biomarker for Post-operative Cognitive Dysfunction in Elderly Patients.
Brief Title: Dexmedetomidine on Postoperative Cognitive Dysfunction and Serum Tau-217 Protein.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Arwa Essam, Assistant Lecturer, Minia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: serum Tau-217 in elderly
Record Dates: First submitted 2024-03-20; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Impairment
Keywords: dexmedetomidine; serum Tau-217 protein; cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Will receive induction of general anesthesia by loading dose of dexmedetomidine (Precedex) 0.6 μg/kg over 10 minutes in a 20 ml micropump, fentanyl in a dose of 1 μg /kg, propofol 1-1.5 mg/kg, and endotracheal intubation will be facilitated by 0.5mg/kg of atracurium and maintenance of anesthesia will be achieved by dexmedetomidine in a dose of 0.3 μg/kg/hr on 50 ml micropump and isoflurane (1-2%) in oxygen-air mixture.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Placebo group (Placebo Comparator): Will receive induction of general anesthesia by infusion of normal saline 20 ml micropump over 10 min, fentanyl in a dose of 1 μg/kg, propofol 1-1.5 mg/kg and endotracheal intubation will be facilitated by 0.5mg/kg of atracurium and maintenance of anesthesia will be achieved by isoflurane (1-2%) in oxygen-air mixture and infusion of 50 ml/hr micropump of normal saline.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — dexmedetomidine effect in preventing postoperative cognitive dysfunction on elderly patients undergoing major surgery guided with serum Tau-217 protein.
  Other Names: precedex
  Arms: Dexmedetomidine group
Other: normal saline — normal saline will be administrated in placebo group
  Arms: Placebo group

SUMMARY:
To assess the effect of Dexmedetomidine on serum Tau-217 protein and its relation to the incidence and severity of postoperative cognitive dysfunction in elderly patients undergoing major surgery under general anesthesia.

DETAILED DESCRIPTION:
to assess the effect of dexmedetomidine on serum Tau-217 protein through measuring serum Tau-217 protein preoperative and postoperative period and comparing the 2 measurements , assessing the cognitive dysfunction in the elderly patients and comparing the correlation between the cognitive dysfunction with serum tau-217 level also assessing the neuroprotective effect of dexmedetomidine on postoperative cognitive dysfunction and its relation with serum Tau-217 level.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 65 years old, both genders, Basal Metabolic Index range 18.5 to less than 35 American Society of Anesthesiologists I - III with Glasgow Coma Scale 14-15 undergoing major surgery under general anesthesia.

Exclusion Criteria:

* Patients will be excluded if they refused the enrollment in our study, Glasgow Coma Scale<14 or if there is severe cardiac, liver or renal disease, patients have Alzehimer's Disease or any of the psychotic diseases, poorly educated patients and if there is any sensitivity to given drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the effect of dexmedetomidine on serum Tau-217 protein value. | 2 years
  estimation of the effect of dexmedetomidine on serum Tau-217 protein in postoperative period.

SECONDARY OUTCOMES:
to evaluate the postoperative cognitive dysfunction using Mini-Mental State Scale in both the placebo and dexmedetomidine group. | 2 years
  evaluation of the postoperative cognitive dysfunction by Mini Mental State Scale as >25 is recorded normal while less than <24 is positive for cognitive dysfunction.

OTHER OUTCOMES:
Heart Rate changes in the intraoperative period after induction of anesthesia and every 10 minutes till the end of surgery and postoperative period after 1 hour and every hour till 6 hours postoperative then every 6 hours | 2 years
  Heart Rate will be measured in beat/min
Mean Arterial Blood Pressure changes in the intraoperative period after induction of anesthesia and every 10 minutes till the end of surgery and postoperative period after 1 hour and every hour till 6 hours postoperative then every 6 hours | 2 years
  Mean Arterial Blood Pressure will be measured in mmHg/min

CONTACTS AND LOCATIONS:
Locations (1):
- Arwa Essam, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thijssen EH, La Joie R, Strom A, Fonseca C, Iaccarino L, Wolf A, Spina S, Allen IE, Cobigo Y, Heuer H, VandeVrede L, Proctor NK, Lago AL, Baker S, Sivasankaran R, Kieloch A, Kinhikar A, Yu L, Valentin MA, Jeromin A, Zetterberg H, Hansson O, Mattsson-Carlgren N, Graham D, Blennow K, Kramer JH, Grinberg LT, Seeley WW, Rosen H, Boeve BF, Miller BL, Teunissen CE, Rabinovici GD, Rojas JC, Dage JL, Boxer AL; Advancing Research and Treatment for Frontotemporal Lobar Degeneration investigators. Plasma phosphorylated tau 217 and phosphorylated tau 181 as biomarkers in Alzheimer's disease and frontotemporal lobar degeneration: a retrospective diagnostic performance study. Lancet Neurol. 2021 Sep;20(9):739-752. doi: 10.1016/S1474-4422(21)00214-3. PMID 34418401
- [Background] McKay TB, Qu J, Liang F, Mueller A, Wiener-Kronish J, Xie Z, Akeju O. Tau as a serum biomarker of delirium after major cardiac surgery: a single centre case-control study. Br J Anaesth. 2022 Jul;129(1):e13-e16. doi: 10.1016/j.bja.2022.04.002. Epub 2022 Apr 22. No abstract available. PMID 35465951
- [Background] Ballweg T, White M, Parker M, Casey C, Bo A, Farahbakhsh Z, Kayser A, Blair A, Lindroth H, Pearce RA, Blennow K, Zetterberg H, Lennertz R, Sanders RD. Association between plasma tau and postoperative delirium incidence and severity: a prospective observational study. Br J Anaesth. 2021 Feb;126(2):458-466. doi: 10.1016/j.bja.2020.08.061. Epub 2020 Nov 20. PMID 33228978
- [Background] Liang F, Baldyga K, Quan Q, Khatri A, Choi S, Wiener-Kronish J, Akeju O, Westover MB, Cody K, Shen Y, Marcantonio ER, Xie Z. Preoperative Plasma Tau-PT217 and Tau-PT181 Are Associated With Postoperative Delirium. Ann Surg. 2023 Jun 1;277(6):e1232-e1238. doi: 10.1097/SLA.0000000000005487. Epub 2022 Jul 6. PMID 35794069
- [Background] Wang W, Ma Y, Liu Y, Wang P, Liu Y. Effects of Dexmedetomidine Anesthesia on Early Postoperative Cognitive Dysfunction in Elderly Patients. ACS Chem Neurosci. 2022 Aug 3;13(15):2309-2314. doi: 10.1021/acschemneuro.2c00173. Epub 2022 Jul 21. PMID 35864562